CLINICAL TRIAL: NCT02068560
Title: The Effect of Gender on Antidiuresis - Evaluated by Graded Low Dose Desmopressin Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GenderDifferences
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-02

CONDITIONS: Gender Difference in V2 Receptor Function in Response to dDAVP Infusion; Nocturia; Nocturnal Enuresis
MeSH Terms: conditions — Nocturia; Nocturnal Enuresis | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dDAVP infusion (Experimental): During the 9 hour study period, the subjects will receive three doses of dDAVP infusion (0.0003micrg/kg, 0.0005micrg/kg, 0.004micrg/kg).
  Interventions: Drug: dDAVP infusion

INTERVENTIONS:
Drug: dDAVP infusion
  Other Names: desmopressin; minirin

SUMMARY:
There is substantial evidence that women throughout life have significantly lower plasma levels of the antidiuretic hormone vasopressin (pAVP) compared to men. The importance of this is not yet fully elucidated, but in relation to the observations of lower pAVP levels, no significant difference in renal response parameters was found. This could be interpreted an increased renal sensitivity in females compared to males. The theory of increased renal sensitivity in females is supported by a few pharmacodynamic studies currently available on this topic. However none of the studies was designed with the purpose of investigate the gender difference.

The aim of this study is to investigate possible gender differences in the renal sensitivity to dDAVP and the effect of age on these differences. This will be done by low dose graded infusion of the synthetic AVP analog dDAVP.

Participants are 80 healthy volunteers equally distributed between four age groups, 8-10 years of age, 16-18 years of age, 25-40 years og age and 65+ years of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Normal clinical examination
* Normal residual urine measurements
* Normal urine dip stick
* Informed consent by participant or legal guardian

Exclusion Criteria:

* Smoking, alcohol or drug abuse
* Conditions of importance to the results (endocrinological, renal or cardial)
* Current or previous history of incontinence, bedwetting or nocturia
* Drug use of importance (diuretics, hormone replacement therapy, birth control pills, desmopressin)
* Pregnancy
* Allergy towards dDAVP/desmopressin

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Urine osmolality | Samples for urine osmolality is measured every half hour throughout the 9 hour study period and measured the following day
Urine Volume | Urine Volume is measured every half hour throughout the 9 hours study period
Plasma dDAVP | Plasma concentrations of the synthetic hormone is measured every 90 minutes for the first 8 hours and every half hour, the last hour of the study period

SECONDARY OUTCOMES:
Plasma sodium | Plasma sodium is measured every 90 minutes throughout the first 8 hours and every half hour in the last hour of the study periode

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark